CLINICAL TRIAL: NCT02321722
Title: The Effect of Colonoscopy on Intralocular Pressure
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Ilan Kent, Medical Doctor, Meir Medical Center
Other Study IDs: MMC-0125-14
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Intraocular Pressure
Keywords: Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Glaucoma is an eye disease that damages the optic nerve, it cause blindness if not diagnosed and treated properly. The major risk factor for the development and progression of glaucoma is increased intraocular pressure. Colonoscopy is one of the most preformed world wide screening exam. It is used to detect colon cancer at its early stages. As part of this examination, the examiner inflates the inspected colon with air in order to increase the colon lumen for better visualization of the colon. As a consequence of the insufflation the intrabdominal pressure increases as well. the increase in intrabdominal pressure could increase intraocular pressure. The aim of this study is to evaluate the intraocular pressure increase while preforming colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age >18.
* Patients referred by a gastroenterologist for a colonoscopy examination.
* Patients the are interested in participating in this study and who are able to sign an informed consent.

Exclusion Criteria:

* Family history of Glaucoma - first degree relatives.
* Patients with known ocular disease, excluding refraction.
* Patients receiving eye pharmacologic treatment.
* Patients with known allergies to Oxybuprocaine Hydrochloride drops.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population are healthy examinees, undergoing routine colonsocopy examination. All have no ocular disese and family history of glucoma.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Increase of Intraocular pressure | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel